CLINICAL TRIAL: NCT05403216
Title: Clinical Value of the Relationship Between Oral Lichen Planus and Autoimmune Thyroid Diseases
Brief Title: Relationship Between Oral Lichen Planus and Autoimmune Thyroid Diseases
Status: Completed | Type: Observational
Sponsor: The Dental Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Qianming Chen, professor, The Dental Hospital of Zhejiang University School of Medicine
Other Study IDs: I20210609
Record Dates: First submitted 2022-03-13; First posted 2022-06-03 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Oral Lichen Planus
MeSH Terms: conditions — Lichen Planus, Oral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsy is the gold standard for the diagnosis of oral lichen planus. Without compromising the diagnosis, we collected oral mucosal tissue from biopsy of oral lichen planus patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- OLP(-): Oral lichen planus (OLP) with negative thyroid antibody group
- OLP(+): OLP with positive thyroid antibody group
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention
  Groups: OLP(+)

SUMMARY:
On the basis of previous studies, a validation cohort will be established to explore the relationship between oral lichen planus and autoimmune thyroid diseases, and a disease efficacy prediction strategy can be formed.

DETAILED DESCRIPTION:
For oral lichen planus patients, the prevalence of Hashimoto's thyroiditis will be investigated and the relationship between levels of anti-TG, anti-TPO antibodies and severity of oral lichen planus will be determined.

Besides, for patients with Hashimoto's thyroiditis, the prevalence of oral lichen planus will be investigated and the relationship between levels of anti-TG, anti-TPO antibodies and severity of oral lichen planus will be determined.

ELIGIBILITY:
Inclusion Criteria:

* OLP patients without systemic disease

Exclusion Criteria:

* OLP patients with severe periodontal disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Oral lichen planus (OLP) patients
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Oral lichen planus (OLP) lesions record | 1 year
  Record changes of lesions based on the symptoms and signs of the oral lichen planus patient.
Level of thyroid function and antibody | 1 year
  The levels of thyroid hormone and thyroid autoantibodies in serum of OLP patients were detected.

CONTACTS AND LOCATIONS:
Overall Officials: Qianming Chen, Dr., Study Chair — Zhejiang University
Locations (1):
- The Stomatology Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No